CLINICAL TRIAL: NCT07078188
Title: The Effect of Discharge Education on PEG Use Given to Palliative Care Patients' Relatives on the Care Burden and Quality of Life of Patients' Relatives
Brief Title: The Effect of PEG Use Education on the Care Burden and Quality of Life of Patients' Relatives
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hicran Yıldız, Prof.Dr., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HYildiz
Record Dates: First submitted 2025-06-15; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Palliative Care; Caregiver; Caregiver Burden of Caregivers; Quality of Life of Caregivers; PEG Training
Keywords: Palliative care; Nutrition; PEG; Caregiver; caregiver burden; Quality of life; PEG training
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Quasi-experimental
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): PEG education
  Interventions: Behavioral: PEG training
- Control (Other)
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: PEG training — The caregivers will be given a general information form, the Caregiver Burden Scale, the Caregiver Stress Index Form, the SF 36 Quality of Life Scale, and the Caregiver Knowledge Scale for Nutrition with Percutaneous Endoscopic Gastrostomy Tube at each meeting (0, 1, and 3 months.). The intervention group will be trained on PEG use before discharge at the first interview.
  Arms: Intervention
Other: Control — The caregivers will be given a general information form, the Caregiver Burden Scale, the Caregiver Stress Index Form, the SF 36 Quality of Life Scale, and the Caregiver Knowledge Scale for Nutrition with Percutaneous Endoscopic Gastrostomy Tube at each meeting (0.,1. ve 3. monts).
  Arms: Control

SUMMARY:
The study was planned to evaluate the effects of discharge training on PEG use given to palliative care patients' relatives on the caregiver burden and quality of life of the relatives.

The main questions that the study aims to answer are as follows:

* How does PEG training given before discharge affect the knowledge level of caregivers on PEG use?
* How does PEG training given before discharge affect the caregiver burden?
* How does PEG training given before discharge affect the caregiver's caregiver stress?
* How does PEG training given before discharge affect the quality of life of the caregivers?

The researchers will compare the PEG training given before discharge with a control group that did not receive training in this regard in order to evaluate the effects of PEG training given before discharge on the caregiver burden, caregiver stress and quality of life of the caregivers. The study will use a general information form, the Caregiver Burden Scale, the Caregiver Stress Index Form, the SF 36 Quality of Life Scale, and the Percutaneous Endoscopic Gastrostomy Tube Nutrition Information Scale for Caregivers.

Participants:

* Face-to-face interviews will be conducted with caregivers at 0, 1, and 3 months.
* The forms used in the study will be filled out at each interview.
* The intervention group will be trained only at the first interview.

ELIGIBILITY:
Inclusion Criteria:

* The caregiver must be over 18 years old
* The caregiver must be willing and able to participate in the study
* The caregiver must be primarily responsible for the patient's care
* The patient they are caring for must be receiving palliative care
* The patient they are caring for must be receiving PEG feeding
* The patient they are caring for must be over 18 years old
* The patient they are caring for must have been diagnosed with stroke at least six months ago
* The caregiver must have a mini mental test score of 25 points or more
* The Beck depression scale score must be under 17 points
* The caregiver must have a score of over 16 points on the Readiness to Provide Care Scale

Exclusion Criteria:

* The caregiver is under the age of 18
* The caregiver is not willing and able to participate in the research
* The caregiver has a physical disability or serious health problem that makes it difficult to provide care
* The patient they are caring for is under the age of 18
* The patient they are caring for has been diagnosed with cancer, endocrine system or GI disease
* The caregiver has a mini mental test score of less than 25
* The Beck depression scale score is 17 points or higher
* The caregiver has scored 16 or lower on the Readiness to Provide Care Scale
* The caregiver has communication problems
* The caregiver has been diagnosed with depression or psychiatric disorder
* The caregiver is receiving psychotherapy/psychological support
* The caregiver is taking antidepressants and/or anxiolytics
* The caregiver has sensory loss related to vision and hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver burden of caregivers | 0th month (1st day), 1st month and 3rd month
  The Caregiver Burden Scale
The quality of life score of the caregivers | 0th month (1st day), 1st month and 3rd month
  The SF 36 Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Yıldız, Prof.Dr., Principal Investigator — Bursa Uludag Unversity
Locations (1):
- Üsküdar State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individuals included in the study were informed that the data obtained would be used and published only within the scope of this study, on condition that their identities remained confidential.